CLINICAL TRIAL: NCT01899781
Title: Prophylactic Antibiotic Treatment for Hand Lacerations Involving Flexor and/or Extensor Tendon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMC-003812-CTIL
Record Dates: First submitted 2013-07-11; First posted 2013-07-15 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Hand Laceration; Tendon Involved; Clean Laceration; No Bone Involved
Keywords: Lacerations; Tendons; Antobiotic
MeSH Terms: conditions — Lacerations | interventions — Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- with antibiotic and without antibiotic (Experimental)
  Interventions: Drug: Antibiotic-Cefamezin

INTERVENTIONS:
Drug: Antibiotic-Cefamezin
  Other Names: Ceforal; Keflex

SUMMARY:
The investigators assume that simple hand lacerations involving flexors or extensors tendons, do not require prophylactic antibiotic treatment to prevent wound infection.

DETAILED DESCRIPTION:
Hand lacerations are divided to "complicated" which involves tendons, nerves, bones, and joints, and "simple" which involves only cutaneous and subcutaneous tissue.

prophylactic antibiotic should not be given in a clean simple lacerations, and should be given when a bone is involve (open fracture). But there is not enough data, weather prophylactic antibiotic treatment should be given when only tendons are involved. The investigators will examine 2 groups of 30 patients each with clean hand lacerations involving tendons. One group will be treated with prophylactic antibiotic and the other wont be treated, randomly. The investigators assume that the rate of wound infection wont be different between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Hand laceration
* Tendon involeved
* Clean laceration
* No bone involved

Exclusion Criteria:

* Pregnant
* Children
* Immunocompremised patients
* "Dirty" lacerations

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
rate of wound infections | 2 years
  signs of wound/tissue infection, levels of WBC, ESR, CRP